CLINICAL TRIAL: NCT03857269
Title: Acupoint Massage and Aromatherapy Intervention in Elderly People With Mild Cognitive Impairment in Nursing Institutions: A Multicenter Clinical Trial
Brief Title: Acupoint Massage and Aromatherapy Intervention in Elderly People With Mild Cognitive Impairment in Nursing Institutions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huan Ding (Other)
Responsible Party: Sponsor-Investigator, Huan Ding, School of Nursing, Nanjing University of Traditional Chinese Medicine, Nanjing University of Traditional Chinese Medicine
Organization: Nanjing University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY2019002
Record Dates: First submitted 2019-02-23; First posted 2019-02-27 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Mild Cognitive Impairment
Keywords: acupressure; Aromatherapy; Nursing Homes; china
MeSH Terms: conditions — Cognitive Dysfunction | interventions — lavender oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acupoint Massage group (Experimental): Choose Chinese medicine acupuncture points： Shenting, Baihui, Sishencong, Diwei, Chengling, Fengchi, Fengfu，Zusanli and Sanyinjiao，32 points per acupressure.32 times per acupoint.Intervention frequency will be monday to saturday per week for 6 months.（n=30）
  Interventions: Other: Acupoint Massage
- Aromatherapy group (Experimental): Make a 5x5cm bag and put a cotton ball in the bag and the bag is clipped to the patient's collar.Dispense 10% lavender essential oil, 2-3 drops a day in cotton balls.Cotton ball replacement daily. Intervention frequency will be monday to saturday per week for 6 months.（n=30）
  Interventions: Other: lavender essential oil
- Acupoint Massage and Aromatherapy group (Experimental): At the same time as the acupressure, the essential oil is applied to the collar and begins to sniff.Intervention frequency will be monday to saturday per week for 6 months.（n=30）
  Interventions: Other: Acupoint Massage and lavender essential oil
- Blank control group (No Intervention): The group selects elderly people with MCI who do not receive intervention after informed.Participate in routine activities of Nursing homes.

INTERVENTIONS:
Other: Acupoint Massage — The operators is trained for two weeks. At 9 o'clock in the morning, the elderly are organized by Nursing home to perform acupressure.Intervention frequency will be monday to saturday per week for 6 months.
  Other Names: AM
  Arms: Acupoint Massage group
Other: lavender essential oil — Modulated by an international aroma therapist,The cotton ball containing essential oil is replaced by the operator at 9 am.Intervention frequency will be monday to saturday per week for 6 months.
  Other Names: EO
  Arms: Aromatherapy group
Other: Acupoint Massage and lavender essential oil — At the same time as the acupressure, patients began to smell the essential oil.Intervention frequency will be monday to saturday per week for 6 months.
  Other Names: AM&EO
  Arms: Acupoint Massage and Aromatherapy group

SUMMARY:
This study aims to investigate and compare the intervention effects of acupressure,aromatherapy,combining acupressure and aromatherapy in elderly with mild cognitive impairment. The investigators hypothesize that (1) Combined intervention can induce greater improvements in the outcome measures than single mode of intervention; (2) the improvement in cognitive functions and other outcomes may differ between the groups.

DETAILED DESCRIPTION:
Background and study aims:

Mild cognitive impairment (MCI) or minor neurocognitive disorder is a syndrome defined as an intermediate stage between cognitively intact and clinically diagnosed dementia. The progression rate from MCI to dementia ranges from 10 to 15% each year, and over 50% of the MCI population will develop into severe cognitive impairment or dementia in 5 years.MCI involves functional decline that may include decrements in engagement in meaningful activities and one's own sense of confidence/mastery, and it is associated with depressive symptoms, poor satisfaction with family communication, and declining physical function. Therefore, early detection of the individuals who manifest MCI and provide appropriate interventions may help reduce the burden of their caregivers and the medical expenses of the health-care system. Previous studies found that acupressure or aromatherapy has emerged as an important therapeutic approach for individuals with MCI. However, the intervention effects of combining acupressure or aromatherapy remain to be determined. Furthermore, whether acupressure and aromatherapy should be administered simultaneously is an important question to pursue. The overall goal of this study is to determine and compare the intervention effects acupressure,aromatherapy, and combining acupressure and aromatherapy in individuals with MCI.

Who can participate? Individuals with MCI (≥60).

What does the study involve? The participants will receive acupressure, aromatherapy, combining acupressure and aromatherapy randomly. Intervention frequency will be 5-6 times per week for 6 months. All participants will received pretreatment test, post treatment test, and a 1-month follow-up test.

What are the possible benefits and risks of participating? The possible benefits include improvement in cognitive, and daily functions. There are no risks for participating.

Where to conduct the study? The investigators anticipate recruiting a total of 120 participants from nursing homes from multiple areas in NanJing,china.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese people aged 60 years or above;
2. the MOCA screening score <26, which was corrected based on educational level (Education time <12, plus one point)
3. ability to perform self-care functions on their own;
4. no confirmed diagnosis of dementia, depression or other psychiatric illnesses which would interfere with cognitive performance;
5. capacity to provide informed consent.

Exclusion Criteria:

1. had a medical history of chronic alcoholism or brain trauma occurred in previous years that could interfere with cognition;
2. had been regular users of medications that could affect cognition;
3. had clinical conditions that contraindicated light to moderate physical exercise；
4. any disabilities preventing participation in the MET or KY conditions (e.g. severe visual or hearing impairment);
5. people with olfactory dysfunction or those who are allergic to lavender；
6. skin is broken, can not be massaged；

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Mini-mental State Examination | Change from baseline in Mini-mental State Examination at month 3 and month 6. To investigate the Intelligence state.
  The table is simple and easy to use, widely used at home and abroad, and is the preferred scale for dementia screening. The scale includes the following seven aspects: time-orientation, location-orientation, immediate memory, attention and computational power, delayed memory, language, and visual space.The total score of the scale ranges from 0-30 points. The test scores are closely related to the cultural level. The normal boundary value is:uneducated people（>17）.primary school education（>20）, and middle high school or above（>24）, indicating good mental state. The higher the total score, the better the situation.
Wechsler Intelligence Scale | Change from baseline in Wechsler Intelligence Scale at month 3 and month 6. To investigate the Memory capacity.
  There are ten aspects of the scale. Consult relevant experts and consult literature, this program selects four aspects: logical memory(0~25), association learning(0~21), picture recall(0~20), and number of memories(0~17).Add the total scores, the higher the score, the better the memory.

SECONDARY OUTCOMES:
Geriatric depression scale | Change from baseline in Geriatric depression scale at month 3 and month 6. To investigate the Functional Activities status.
  Dedicated to screening for depression in the elderly. The most suitable feelings for the elderly in the past week were evaluated. The scale has a total of thirty entries, including the following symptoms: low mood, reduced activity, irritability, retreat from painful thoughts, negative scores on past, present and future.The total score is 0-10 points, which is normal; 11-20 points, mild depression; 21-30 minutes, moderate to severe depression.
Pittsburgh sleep quality index | Change from baseline in Pittsburgh sleep quality index at month 3 and month 6. To investigate the Functional Activities status.
  PSQI was used to assess the quality of sleep in the last month of the test. It consists of 19 self-evaluations and 5 other evaluation items. The 19th self-evaluation item and 5 other evaluation items do not participate in the scoring. Only 18 self-evaluation items participating in the scoring are introduced here. 18 items are composed of 7 components, each component is scored according to o~3 level, and the accumulated components are scored as PSQI total score, and the total score range is 0~2l. The higher the score, the worse the sleep quality. It takes 5 to 10 minutes for the subject to complete the test.

CONTACTS AND LOCATIONS:
Overall Officials: Huan Ding, Principal Investigator — School of Nursing, Nanjing University of Traditional Chinese Medicine
Locations (1):
- Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China